CLINICAL TRIAL: NCT05689723
Title: The Effect of Spinal Manipulation on Hip Extension Strength and Jump Height, A Double Blind Randomized Control Trial
Brief Title: The Effect of Spinal Manipulation on Hip Extension Strength and Jump Height
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Messiah College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Bergmann
Record Dates: First submitted 2022-10-03; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-10

CONDITIONS: Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manipulation (Experimental): Left and right sidelyiing gaping high velocity low amplitude thrust mobilization
  Interventions: Procedure: Lumbar manipulation
- Sham Manipulation (Sham Comparator): The experimenter holds both knees with one arm while placing their opposite hand on the participant's lumbar spine. The experimenter performs 1 min of ﬂexion and extension PROM without reaching physiological end range in either direction of movement. This is repeated with the subject in left sidelying.
  Interventions: Procedure: Sham Manipulation

INTERVENTIONS:
Procedure: Lumbar manipulation — Left and right sidelyiing gaping high velocity low amplitude thrust mobilization
  Arms: Manipulation
Procedure: Sham Manipulation — The experimenter holds both knees with one arm while placing their opposite hand on the participant's lumbar spine. The experimenter performs 1 min of ﬂexion and extension PROM without reaching physiological end range in either direction of movement. This is repeated with the subject in left sidelying.
  Arms: Sham Manipulation

SUMMARY:
The purpose of this study is to study the effects of lumbar manipulation on hip extension strength and jump height in healthy subjects.

Procedures to be followed: First, the subject will be asked to complete a medical history form. Then they will be instructed on the procedure for strength and jump testing. Next, range of motion of the low back will be measured. Then hip strength will be measured using a digital handheld measurement tool. The subject will then be asked to jump as high as they can on a floor mat. The subject will then receive a sealed envelope indicating the intervention they will to receive, either the manipulation or a fake manipulation. Instructions will be provided, and the subject will be positioned on a treatment table to receive the intervention. At this point, they will either receive the manipulation or fake manipulation on the right and left side. An immediate re-test of hip strength will be taken, and the subject will again jump as high as they can on a floor mat. Follow-up measures of these tests will be completed again 20 minutes after the intervention is given.

DETAILED DESCRIPTION:
The participant will complete a medical history form and undergo a brief active range of motion screen of the lumbar spine. The participant will complete a hip strength test utilizing the microFET 2 Manual Muscle Tester Hand Held Dynamometer. The participant will then jump as high as they can on the Just Jump System. A sealed envelope indicating the intervention to be received will be given to the participant. An investigator blinded to the pre and post-measures will open the envelope indicating the intervention to be performed. The participant will be blinded to which intervention group they are categorized to. The participant will be positioned on a high-low treatment table to receive the assigned intervention, either intervention 1 (thrust mobilization) or 2 (sham mobilization). The participant will either receive the thrust-mobilization or sham mobilization up to 2 times on the left and right side. An immediate re-test of hip strength will be conducted followed by performing the same three jumps. Follow-up measures at 20 minutes post-intervention will be performed.

Intervention for the Thrust-mobilization Group The intervention group will receive passive spinal rotational grade V mobilization, based on Maitland's approach. The intervention will be performed with the subject in right sidelying and left sidelying. The operator's palpating hand is placed over the L2-3 intervertebral space, and the other hand bends both legs of the participant up to the range at which the L2-3 midposition is found. The participant is then asked to straighten the lower leg and hook the upper leg over it with the upper leg's knee positioned over the side of the plinth. While the lower component is kept still, the participant's trunk is rotated until the hip starts to lift off from the plinth. The bottom hand and uppermost hand rest under a pillow and the chest wall, respectively. With the starting position settled, the operator stands behind the participant, takes up the slack within the spine and then provides a grade V mobilization while stabilizing the uppermost shoulder.

Intervention for the Sham Group Subjects are positioned in right sidelying. The experimenter holds both knees with one arm while placing their opposite hand on the participant's lumbar spine. The experimenter performs 1 min of ﬂexion and extension PROM without reaching physiological end range in either direction of movement. This is repeated with the subject in left sidelying.

Double Blind: The subjects will not know what intervention they are receiving - same generic script is provided. One Investigator is performing all pre and post-tests without knowledge of intervention, the other investigator is opening the envelope and providing the intervention behind a screen without knowledge of test results. This investigator will record the subjects assigned # and which intervention they received. Investigators will record data on spreadsheet separately.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 30
* able to read and write in English and clearly understand the informed consent.

Exclusion Criteria:

* currently have low back pain
* pregnant or may be pregnant
* previously diagnosed with spondylolisthesis, a herniated disc, or have signs and symptoms of nerve root compression
* history of spine surgery
* history of cancer, compression fracture, osteoporosis, osteopenia, or a history of systemic, connective tissue, or neurological disease,
* pain with the pre-manipulative hold
* positive findings on medical history form, or physical exam,
* presence of anxiety during the procedure

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in hip extension strength | immediately post instervention and 20 minutes post
  microFET 2 Manual Muscle Tester Hand Held Dynamometer

SECONDARY OUTCOMES:
Change in jump height | immediately post instervention and 20 minutes post
  Just Jump System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sueki DG, Cleland JA, Wainner RS. A regional interdependence model of musculoskeletal dysfunction: research, mechanisms, and clinical implications. J Man Manip Ther. 2013 May;21(2):90-102. doi: 10.1179/2042618612Y.0000000027. PMID 24421619
- [Background] Wainner RS, Whitman JM, Cleland JA, Flynn TW. Regional interdependence: a musculoskeletal examination model whose time has come. J Orthop Sports Phys Ther. 2007 Nov;37(11):658-60. doi: 10.2519/jospt.2007.0110. No abstract available. PMID 18057674
- [Background] Mintken PE, McDevitt AW, Cleland JA, Boyles RE, Beardslee AR, Burns SA, Haberl MD, Hinrichs LA, Michener LA. Cervicothoracic Manual Therapy Plus Exercise Therapy Versus Exercise Therapy Alone in the Management of Individuals With Shoulder Pain: A Multicenter Randomized Controlled Trial. J Orthop Sports Phys Ther. 2016 Aug;46(8):617-28. doi: 10.2519/jospt.2016.6319. PMID 27477473
- [Background] McDevitt A, Young J, Mintken P, Cleland J. Regional interdependence and manual therapy directed at the thoracic spine. J Man Manip Ther. 2015 Jul;23(3):139-46. doi: 10.1179/2042618615Y.0000000005. PMID 26309384
- [Background] Bergman GJ, Winter JC, van Tulder MW, Meyboom-de Jong B, Postema K, van der Heijden GJ. Manipulative therapy in addition to usual medical care accelerates recovery of shoulder complaints at higher costs: economic outcomes of a randomized trial. BMC Musculoskelet Disord. 2010 Sep 6;11:200. doi: 10.1186/1471-2474-11-200. PMID 20819223
- [Background] Stupar M, Cote P, French MR, Hawker GA. The association between low back pain and osteoarthritis of the hip and knee: a population-based cohort study. J Manipulative Physiol Ther. 2010 Jun;33(5):349-54. doi: 10.1016/j.jmpt.2010.05.008. PMID 20605553
- [Background] Pickar JG. Neurophysiological effects of spinal manipulation. Spine J. 2002 Sep-Oct;2(5):357-71. doi: 10.1016/s1529-9430(02)00400-x. PMID 14589467
- [Background] Espi-Lopez GV, Arnal-Gomez A, Balasch-Bernat M, Ingles M. Effectiveness of Manual Therapy Combined With Physical Therapy in Treatment of Patellofemoral Pain Syndrome: Systematic Review. J Chiropr Med. 2017 Jun;16(2):139-146. doi: 10.1016/j.jcm.2016.10.003. Epub 2016 Nov 22. PMID 28559754
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Ingersoll CD. Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther. 2009 Aug;14(4):415-20. doi: 10.1016/j.math.2008.06.005. Epub 2008 Sep 20. PMID 18805726
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Kerrigan DC, Fan X, Ingersoll CD. Lumbopelvic joint manipulation and quadriceps activation of people with patellofemoral pain syndrome. J Athl Train. 2012 Jan-Feb;47(1):24-31. doi: 10.4085/1062-6050-47.1.24. PMID 22488227
- [Background] Sanders GD, Nitz AJ, Abel MG, Symons TB, Shapiro R, Black WS, Yates JW. Effects of Lumbosacral Manipulation on Isokinetic Strength of the Knee Extensors and Flexors in Healthy Subjects: A Randomized, Controlled, Single-Blind Crossover Trial. J Chiropr Med. 2015 Dec;14(4):240-8. doi: 10.1016/j.jcm.2015.08.002. Epub 2015 Nov 6. PMID 26793035
- [Background] Yuen TS, Lam PY, Lau MY, Siu WL, Yu KM, Lo CN, Ng J. Changes in Lower Limb Strength and Function Following Lumbar Spinal Mobilization. J Manipulative Physiol Ther. 2017 Oct;40(8):587-596. doi: 10.1016/j.jmpt.2017.07.003. PMID 29187310
- [Background] Botelho MB, Alvarenga BAP, Molina N, Ribas M, Baptista AF. Spinal Manipulative Therapy and Sports Performance Enhancement: A Systematic Review. J Manipulative Physiol Ther. 2017 Sep;40(7):535-543. doi: 10.1016/j.jmpt.2017.03.014. PMID 29191288
- [Background] Sandell J, Palmgren PJ, Bjorndahl L. Effect of chiropractic treatment on hip extension ability and running velocity among young male running athletes. J Chiropr Med. 2008 Jun;7(2):39-47. doi: 10.1016/j.jcme.2008.02.003. PMID 19674719